CLINICAL TRIAL: NCT00475007
Title: A Prospective, Randomized, Controlled Multicenter Clinical Trial to Evaluate the Safety and Effectiveness of the IBV® Valve System for the Treatment of Severe Emphysema
Brief Title: Clinical Trial to Evaluate the Safety and Effectiveness of the IBV® Valve System for the Treatment of Severe Emphysema
Acronym: IBV®Valve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPR-01377
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2017-11

CONDITIONS: Emphysema; COPD
Keywords: Emphysema; IBV® Valve; COPD; Shortness of Breath; Spiration
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): The experimental group will have an investigational medical device implanted in their lungs with an instrument known as a bronchoscope. This procedure is done without an incision
  Interventions: Device: IBV® Valve System
- 2 (Sham Comparator): The sham comparator group will be tested, treated and followed in an identical manner as the experimental group, except that no valves will be placed during the diagnostic bronchoscopy, the sham procedure.
  Interventions: Device: IBV® Valve System

INTERVENTIONS:
Device: IBV® Valve System — The IBV Valve is a small, umbrella shaped device designed to redirect airflow to healthier areas of the lungs. It is implanted without incisions using a bronchoscope.

SUMMARY:
This trial is for men and women between the ages of 40 and 74 who have a confirmed diagnosis of emphysema. The objective of the trial is to determine the safety and effectiveness of the IBV Valve at redirecting airflow from diseased portions of the lung to healthier areas to achieve improvement in disease-related health status.

DETAILED DESCRIPTION:
The IBV Valve Trial is a multi-center clinical trial evaluating the IBV Valve System, a non-surgical treatment for patients with emphysema. The IBV Valve System does not require traditional surgery or surgical incisions. The valves are placed during a bronchoscopic procedure. The IBV Valve System is designed to redirect airflow from diseased portions of the lung to healthier areas to achieve improvement in disease-related health status. Although the valves are intended to be permanent, they are designed to be removed if necessary.

The IBV Valve Trial is a randomized, blinded trial. This means that participants are divided into two groups but do not know to which group they have been assigned.

The IBV Valve Treatment Group receives valves, and the Control Group does not. A random selection process decides the group assignments (participants will not be able to choose their group). In the trial, everyone will have a 50 percent chance (similar to a coin toss) to be assigned to one group or the other.

All Participants in this Clinical Trial will:

Receive a diagnostic bronchoscopy that will allow an expert in lung health to evaluate their lungs.

Be under the care of a highly qualified lung doctor for the entire time they are in the trial, regardless of whether they are in the Treatment Group or the Control Group.

Receive regular periodic check-ups and health assessments throughout the 6 month trial period.

The procedure, all testing, and doctor visits are provided at no cost to participants of both the IBV Valve Treatment Group and the Control Group.

At the completion of their 6-month visit, participants will be told if they were assigned to the Treatment Group or the Control Group. If participants were assigned to the group that did not receive valves (the Control Group), they will be given the option to be re-evaluated by the clinical trial doctor, to determine if they can have valve treatment.

ELIGIBILITY:
Inclusion Criteria:

* Candidates have mostly upper lobe, severe emphysema.
* Must be able to participate in standard exercise testing.
* Willing to abstain from cigarette smoking for 4 months prior and during the entire trial.
* Willing to participate in a randomized, blinded study and complete the required follow-up visits during the study period.
* Willing to participate in multiple visits to a medical center for health assessment tests.
* Willing to have a minimum of one overnight stay in the hospital.

Exclusion Criteria:

* Evidence of another co-existing major medical disease.
* Unable to tolerate, flexible bronchoscopy procedures.
* Active asthma, chronic bronchitis.
* Diffuse emphysema pattern, alpha 1-antitrypsin deficiency.
* Has had prior lung volume reduction surgery.

Ages: 40 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2007-09 (Actual); Primary Completion 2011-02 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Difference between responder rates of the treatment & control groups, responders defined as subjects with clinically meaningful improvements in disease-related health status (SGRQ) & regional lung volume changes as measured by quantitative CT scan. | 6 months

SECONDARY OUTCOMES:
The difference between average 6 minute walk test results for treatment & control groups. | 6 months

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Kaiser Permanente Medical Center, Los Angeles, California
  - University of California Los Angeles (UCLA), Los Angeles, California
  - Mission Internal Medicine Group, Mission Viejo, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Diego, San Diego, California
  - National Jewish Medical & Research Center, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Emory HealthCare, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - Alexian Brothers Hospital Network, Elk Grove Village, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Louisville, Louisville, Kentucky
  - Pulmonary and Critical Care Associates of Baltimore, Baltimore, Maryland
  - Health Partners Research Foundation/Regions Hospital, Saint Paul, Minnesota
  - Pulmonary and Allergy Associates, Summit, New Jersey
  - Mount Sinai School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - Akron General Medical Center, Akron, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oklahoma State University, Tulsa, Oklahoma
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Health Science Center, San Antonio, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
  - Franciscan Research Center, Tacoma, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Wood DE, Nader DA, Springmeyer SC, Elstad MR, Coxson HO, Chan A, Rai NS, Mularski RA, Cooper CB, Wise RA, Jones PW, Mehta AC, Gonzalez X, Sterman DH; IBV Valve Trial Research Team. The IBV Valve trial: a multicenter, randomized, double-blind trial of endobronchial therapy for severe emphysema. J Bronchology Interv Pulmonol. 2014 Oct;21(4):288-97. doi: 10.1097/LBR.0000000000000110. PMID 25321447